CLINICAL TRIAL: NCT06103383
Title: Second Phase of the Pilot Study for Obtaining Mature Oocytes by in Vitro Maturation in Oocyte-donor Women
Acronym: MIVODON-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2109-VLC-083-EB
Record Dates: First submitted 2023-10-23; First posted 2023-10-26 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Infertility, Female; Oocyte Maturation
Keywords: IN VITRO MATURATION; OOCYTE ACTIVATION; FOLLICULAR PUNCTURE; hMG-HP; OOCYTE DONNORS
MeSH Terms: conditions — Infertility, Female | interventions — In Vitro Oocyte Maturation Techniques

STUDY DESIGN:
Intervention Model Description: Prospective, observational, single-center, prospective cohort pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donors with history of optimal ovarian response (Experimental): IVIRMA Valencia donors between the ages of 18-35 years old, with normal ovarian function, with a history of optimal ovarian response (at least 10 total oocytes and/or 8 MII) and who have already completed all their donation cycles allowed by law.
  Interventions: Drug: Controlled ovarian stimuation; Procedure: Oocyte pick up; Procedure: Oocyte in vitro maturation; Procedure: Oocyte in vitro activation

INTERVENTIONS:
Drug: Controlled ovarian stimuation — 3 days stimullation protocol using hMG-HP
Procedure: Oocyte pick up — Surgical oocyte pick up without triggering
Procedure: Oocyte in vitro maturation — In vitro maturation procedure
Procedure: Oocyte in vitro activation — In vitro oocyte activation procedure

SUMMARY:
In vitro maturation (IVM) is a technique for obtaining potentially fertilizable oocytes from immature oocytes. An oocyte must be mature both nuclearly and cytoplasmically in order to be competent in the reproductive process. Nuclear maturation involves an oocyte in metaphase II stage and is easily evaluated for its morphology. However, cytoplasmic maturation can only be evaluated by in vitro fertilization of that oocyte. A mature nuclear and cytoplasmic oocyte is the one capable of producing a viable embryo. This study aims to optimize the in vitro maturation (IVM) technique to achieve nuclear mature oocytes, i.e., to mature the oocytes up to the metaphase II stage. In addition, an artificial oocyte activation (AOA) will be carried out to check the cytoplasmic maturation of the oocytes, avoiding the generation of potentially viable embryos.

This study corresponds to a second phase of the pilot study for the development of this technique in our IVF laboratory. We will use all we have learned in the first phase, as well as the experience acquired, to advance in the optimization of this protocol.

The correct functioning of this IVM technique would mean a reduction in the costs of ovarian stimulation treatments, as lower doses and shorter stimulation times are required, which implies lower risks for women derived from the medication and less stress for them.

ELIGIBILITY:
-Inclusion criteria:

Women between 18-35 years old who have belonged to the egg donation program. Donors who agree to participate in the study after informing and signing the Informed Consent.

Documented previous good response to ovarian stimulation (at least 10 total oocytes and/or 8 MII).

Donors with at least one previous donation cycle, in which all oocytes obtained were freshly fertilized.

Donors who have already done all their donation cycles allowed by law. No personal or family history of interest.

From the medical point of view:

Body mass index between 18-25 kg/m2. Normal uterus and ovaries, without organic pathology. No polycystic ovaries Antral follicle count (AFC) >12 in the sum of the two ovaries on day 2-3 of the menstrual cycle. Normal karyotype Negative screening for infectious diseases (Hepatitis B virus, Hepatitis C virus, Human Immunodeficiency Virus and Syphilis). General analysis with hemogram, hemostasis and biochemistry with parameters within normality.

-Exclusion criteria:

Any systemic or metabolic disorder that contraindicates the use of gonadotropins.

Any medical condition that implies non-inclusion in the oocyte donation program.

Taking hormonal contraceptives within the last 3 months.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Oocyte in-vitro maturation | 1 YEAR
  To evaluate the rate of potentially competent oocytes (after the in vitro maturation).
Oocyte activation | 1 YEAR
  To evaluate the rate of potentially competent oocytes after oocyte activation process.

SECONDARY OUTCOMES:
Oocyte recovery rate | 1 year
  To evaluate Oocyte recovery rate per punctured follicle
In vitro nuclear maturation rate | 1 year
  To evaluate In vitro nuclear maturation rate per punctured follicle
Artificial oocyte activation rate. | 1 year
  To evaluateArtificial oocyte activation rate. per punctured follicle

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Bosch, PhD, Principal Investigator — IVIRMA Valencia
Locations (1):
- Ivi Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No